CLINICAL TRIAL: NCT04040777
Title: Cardiometabolic Risk Factors Registry
Acronym: CARFARE
Status: Recruiting | Type: Observational
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Coordinator of Clinical Research Department, Austral University, Argentina
Other Study IDs: 19-044
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Atherosclerosis; Metabolic Syndrome; Diabetes; Cardiovascular Risk Factor; Cardiovascular Diseases; Obesity
Keywords: Subclinical Atherosclerosis; Metabolic Syndrome; Primary Prevention
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome; Diabetes Mellitus; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CARFARE (CARDIOMETABOLIC RISK FACTORS REGISTRY) is a registry done in the context of a cardiovascular primary prevention program of the Cardiometabolic Unit Officia of the Cardiology Department of the Austral University Hospital. The structured and sequential evaluation include measurement of anthropometric parameters (body mass index, BMI), laboratory with metabolic profile, baseline electrocardiogram, blood pressure (BP) measurement, arterial stiffness, subclinical atherosclerosis screening in the carotid and ileo-femoral territories using echo-doppler, echocardiogram, and ergometry test.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.

Exclusion Criteria:

* Previous cardiovascular and/or cerebrovascular event
* stable chronic angina
* advanced chronic kidney disease (Stage IV or V)
* cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary prevention population. Most of the population are low and moderate cardiovascular risk.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 5 years
  Inicidence of myocardial infarction, stroke, unstable angina or acute heart failure
Mortality rate | 5 years
  Death due to MACE or other causes

CONTACTS AND LOCATIONS:
Overall Officials: Maximo A Schiavone, MD, Principal Investigator — Austral University, Argentina; Sergio Gonzalez, MD, Study Director — Austral University, Argentina
Locations (1):
- Hospital Universitario Austral, Pilar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No